CLINICAL TRIAL: NCT06353269
Title: Adherence to Vaginal Estrogen Therapy in Hypoestrogenic Women With Recurrent Urinary Tract Infections
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Charlotte Ter Haar, Resident Physician, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4255
Record Dates: First submitted 2024-02-28; First posted 2024-04-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Urinary Tract Infection; Hypoestrogenism
Keywords: vaginal estrogen
MeSH Terms: conditions — Urinary Tract Infections | interventions — Estradiol; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Estrogen cream (Experimental): Participants in this arm will receive the vaginal estrogen cream (Estrace 0.01%) for treatment. Participants will apply 0.5gm twice per week for the duration of the study.
  Interventions: Drug: Estrace 0.01% Vaginal Cream
- Estrogen tablet (Experimental): Participants in this arm will receive the vaginal estrogen tablets (Vagifem) for treatment. Participants will place one tablet (10 mcg) into the vagina twice per week for the duration of the study.
  Interventions: Drug: Vagifem
- Estrogen drug-eluting ring (Experimental): Participants in this arm will receive the vaginal estrogen drug-eluting ring (Estring) for treatment. Participants will have the ring placed by a provider at their clinical visit. The ring will be exchanged every 12 weeks.
  Interventions: Drug: Estring Vaginal Product

INTERVENTIONS:
Drug: Estring Vaginal Product — estradiol vaginal ring, exchanged every 12 weeks
  Arms: Estrogen drug-eluting ring
Drug: Vagifem — vaginal estrogen tablet, used twice per week
  Arms: Estrogen tablet
Drug: Estrace 0.01% Vaginal Cream — vaginal estrogen cream, used twice per week
  Arms: Estrogen cream

SUMMARY:
* The goal of this clinical trial is to learn about medication adherence to difference types of vaginal estrogen in women with low levels of estrogen (for example, post-menopausal women) who have recurrent urinary tract infections. Medication adherence means whether patients take their medicine as prescribed.
* Another goal of the study is to learn about changes to the skin of the vagina before and after estrogen treatment, using a specialized imaging modality called optical coherence tomography, which is similar to receiving an ultrasound.
* A third goal of the study is to learn about changes to the microbiome (all the bacteria that naturally live in our bodies) before and after treatment with vaginal estrogen. The researchers will be looking specifically at the microbiome in the urine and the vagina.

Participants will be assigned by chance (like the flip of a coin) to receive one of three possible vaginal estrogen treatments - cream, tablets, or drug-eluting ring.

* The main study tests and procedures include an initial visit in which the researchers will collect baseline information about participants and have participants complete a series of questionnaires.
* There will then be 3 and 6 month follow-ups in which the researchers will have participants complete additional questionnaires and the researchers also assess whether participants are using the vaginal estrogen treatment that you were prescribed.

If a participant is part of the microbiome cohort, they will also be asked to do the following:

* a baseline visit in which urinary and vaginal specimens are collected to assess their baseline microbiome. The vaginal specimen collection will involve a q-tip swab inside the vagina; it is similar to a pap smear.
* Finally, participants will have an imaging modality performed on their vagina called optical coherence tomography, which allows the researchers to assess the thickness of the vaginal walls and the blood vessel density. This imaging modality involves the insertion of a thin probe into the vagina to obtain the images of the vaginal wall.
* These tests will then be repeated at 6 months to assess if vaginal estrogen treatment causes changes to the vagina.

ELIGIBILITY:
Inclusion Criteria:

* female, at least 18 years old with diagnosis of hypoestrogenism (defined by post-menopausal status of 12 months or more of amenorrhea, history of bilateral salpingo-oophorectomy) AND recurrent UTI as defined by greater than or equal to 3 in 1 year or 2 in 6 months by positive urine culture or clinically suspected UTI)

Exclusion Criteria:

* Have a known etiology of infections (urologic stones, fistulas, fecal incontinence, catheterization, or poorly controlled diabetes - Hgb A1C cutoff of 8)
* Contraindication to vaginal estrogen (actively treated estrogen-sensitive tumor, allergies to medication formulation, inability to apply or place vaginal estrogen of any modality)
* Suspected mesh complications or voiding problems from pelvic reconstructive surgery
* Short vaginal length (less than 7cm) or poor dexterity or mobility that may prevent use of estrogen ring
* Do not speak English
* For the nested cohort only - patients currently using vaginal estrogen greater than 2x per month

Deferral criteria:

* Undiagnosed hematuria or vaginal bleeding; however enrollment may proceed after negative workup for malignancy
* Remote history of estrogen-sensitive tumor: enrollment allowed after approval by oncologist or primary care physician

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Adherence to vaginal estrogen treatment | 6 month follow-up visit
  The primary outcome will be the adherence to vaginal estrogen treatment at the 6 month follow-up visit. The 6 month follow-up visit will be the endpoint of the study. The investigators will consider both subjective, patient-reported adherence at 6 months, as well as objective data - tube weight for the estrogen cream, number of tablets left for the estrogen tables, and presence or absence of drug-eluting ring on physical exam for the estrogen ring.

SECONDARY OUTCOMES:
UTI rates | the 6 month duration of the study
  number of culture-proven urinary tract infections
validated patient questionnaire - Urinary Distress Inventory Short Form (UDI-6) | Questionnaires will be collected at the baseline visit, 3 month follow-up and 6 month follow-up
  Urinary Distress Inventory Short Form (UDI-6) - six questions, scored from 0 (not at all) to 3 (greatly), with higher scores indicating more distress from urinary symptoms.
validated patient questionnaires - UTI Symptoms Assessment Questionnaire (UTISA) | Questionnaires will be collected at the baseline visit, 3 month follow-up and 6 month follow-up
  UTI Symptoms Assessment Questionnaire (UTISA) - 15 questions, rated from 0 (did not have/not at all) to 3 (severe/a lot), with higher scores indicating a more symptomatic UTI
validated patient questionnaires - Treatment Satisfaction with Medications Questionnaire (SATMED-Q) | Questionnaires will be collected at the baseline visit, 3 month follow-up and 6 month follow-up
  Treatment Satisfaction with Medications Questionnaire (SATMED-Q) - 17 questions, scored from 0 (not at all) to 4 (very much), with higher scores indicating greater satisfaction with medical treatment.
validated patient questionnaires - Patient Global Impression of Improvement Questionnaire (PGI-I) | Questionnaires will be collected at the baseline visit, 3 month follow-up and 6 month follow-up
  Patient Global Impression of Improvement Questionnaire (PGI-I) - one-question with scores from 1 (very much better) to 7 (very much worse0, with higher scores indicating a worsening in symptoms after treatment.
validated patient questionnaires - Medication Adherence Report Scale (MARS-5) | Questionnaires will be collected at the baseline visit, 3 month follow-up and 6 month follow-up
  Medication Adherence Report Scale (MARS-5) - 5 questions, rated from 1 (always) to 5 (never), with a higher score indicating lower medication adherence.
optical coherence tomography measurements for nested OCT cohort - vaginal epithelial thickness | baseline and 6 month follow-up visits
  changes to vaginal epithelial thickness (VET) before and after treatment as measured by vaginal optical coherence tomography (OCT).
optical coherence tomography measurements for nested OCT cohort - blood vessel density | baseline and 6 month follow-up visits
  changes to blood vessel density (BVD) before and after treatment as measured by vaginal optical coherence tomography (OCT).
Vaginal health index for nested microbiome cohort | baseline and 6 month follow-up visits
  vaginal health index (VHI) before and after treatment - The Vaginal Health Index Score is a clinical tool that, by evaluating 5 parameters (vaginal elasticity, vaginal secretions, pH, epithelial mucous membrane, vaginal hydration), allows to obtain a final score defining the degree of atrophy in the genitourinary tract by assigning a single score to each parameter. Total score ranges from 5 to 25, with lower scores corresponding to greater urogenital atrophy
Vaginal maturation index for nested microbiome cohort | baseline and 6 month follow-up visits
  vaginal maturation index (VMI) before and after treatment - microscopic evaluation of the ratio of vaginal epithelial cells (parabasal, intermediate and superficial)
Urologic microbiome results for nested microbiome cohort | baseline and 6 month follow-up visits
  Urologic microbiome before and after treatment (Lactobacillus abundance processed by Zymo analysis).
Vaginal microbiome results for nested microbiome cohort | baseline and 6 month follow-up visits
  Vaginal microbiome before and after treatment (Lactobacillus abundance processed by Zymo analysis).

CONTACTS AND LOCATIONS:
Overall Officials: CHARLOTTE TER HAAR, MD, Principal Investigator — University of California, Irvine; Olivia Chang, MD, Study Director — University of California, Irvine
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foxman B. Epidemiology of urinary tract infections: incidence, morbidity, and economic costs. Am J Med. 2002 Jul 8;113 Suppl 1A:5S-13S. doi: 10.1016/s0002-9343(02)01054-9. PMID 12113866
- [Background] Tan-Kim J, Shah NM, Do D, Menefee SA. Efficacy of vaginal estrogen for recurrent urinary tract infection prevention in hypoestrogenic women. Am J Obstet Gynecol. 2023 Aug;229(2):143.e1-143.e9. doi: 10.1016/j.ajog.2023.05.002. Epub 2023 May 11. PMID 37178856
- [Background] Perrotta C, Aznar M, Mejia R, Albert X, Ng CW. Oestrogens for preventing recurrent urinary tract infection in postmenopausal women. Obstet Gynecol. 2008 Sep;112(3):689-90. doi: 10.1097/AOG.0b013e318185f7a5. No abstract available. PMID 18757671
- [Background] Brubaker L, Carberry C, Nardos R, Carter-Brooks C, Lowder JL. American Urogynecologic Society Best-Practice Statement: Recurrent Urinary Tract Infection in Adult Women. Female Pelvic Med Reconstr Surg. 2018 Sep/Oct;24(5):321-335. doi: 10.1097/SPV.0000000000000550. No abstract available. PMID 29369839
- [Background] Raz R, Stamm WE. A controlled trial of intravaginal estriol in postmenopausal women with recurrent urinary tract infections. N Engl J Med. 1993 Sep 9;329(11):753-6. doi: 10.1056/NEJM199309093291102. PMID 8350884
- [Background] Eriksen B. A randomized, open, parallel-group study on the preventive effect of an estradiol-releasing vaginal ring (Estring) on recurrent urinary tract infections in postmenopausal women. Am J Obstet Gynecol. 1999 May;180(5):1072-9. doi: 10.1016/s0002-9378(99)70597-1. PMID 10329858
- [Background] Portman D, Shulman L, Yeaw J, Zeng S, Uzoigwe C, Maamari R, Iyer NN. One-year treatment persistence with local estrogen therapy in postmenopausal women diagnosed as having vaginal atrophy. Menopause. 2015 Nov;22(11):1197-203. doi: 10.1097/GME.0000000000000465. PMID 25944522
- [Background] Minkin MJ, Maamari R, Reiter S. Improved compliance and patient satisfaction with estradiol vaginal tablets in postmenopausal women previously treated with another local estrogen therapy. Int J Womens Health. 2013;5:133-9. doi: 10.2147/IJWH.S41897. Epub 2013 Mar 15. PMID 23526171
- [Background] Weissmann-Brenner A, Bayevsky T, Yoles I. Compliance to vaginal treatment-tablets versus cream: a retrospective 9 years study. Menopause. 2017 Jan;24(1):73-76. doi: 10.1097/GME.0000000000000729. PMID 27648663
- [Background] Rioux JE, Devlin C, Gelfand MM, Steinberg WM, Hepburn DS. 17beta-estradiol vaginal tablet versus conjugated equine estrogen vaginal cream to relieve menopausal atrophic vaginitis. Menopause. 2000 May-Jun;7(3):156-61. doi: 10.1097/00042192-200007030-00005. PMID 10810960